CLINICAL TRIAL: NCT03512678
Title: A Multi-Centric Evaluation of a Device for Automated Malaria Microscopy (EasyScan Go)
Brief Title: Evaluation of a Digital Microscope for Malaria
Acronym: EasyScanGo
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: MAL18002
Record Dates: First submitted 2018-04-18; First posted 2018-05-01 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection from finger-prick (maximum 150-200 µL), which will be used to prepare slides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Light microscopy, which is based on century-old technology, remains a key indicator in drug efficacy testing performed in the context of clinical trials for monitoring existing antimalarial drugs or in the context of regulatory clinical trials for registration of new drugs. It is one of the main diagnostic methods for malaria diagnosis in general, as in an ideal setting it can provide low-cost accurate diagnosis, determine the density of parasites in the blood, and accurately differentiate between different malaria parasite species, characteristics vital to the implementation of global plans for drug efficacy monitoring. Malaria rapid tests (RDTs), while useful for rapid diagnosis and case management, do not provide information on the parasite density nor the species differentiation necessary for research and drug efficacy assessment. Microscopy therefore retains key advantages over a number of newer technologies, but its reliability is severely impeded by dependence on high technical competence of the human operators as well as availability of high quality equipment and reagents. Recent studies have demonstrated frequent poor specificity and sensitivity associated with manual microscopy diagnostics in operational conditions. These drawbacks constitute a major limiting factor to effective monitoring and preservation of vital anti-malarial medicines.

Advances in digital microscopy performance and affordability have now opened the door to potentially significant improvements in the performance of malaria microscopy, overcoming serious deficiencies in current drug efficacy assessment, and more broadly in malaria diagnosis and management. Global Good (GG)/Intellectual Ventures Laboratory (IVL) sponsored by the Global Good Fund, has developed a microscope prototype consisting of low cost components to scan and capture images from Giemsa-stained thick blood films on slides. The captured images are analyzed with custom image analysis software developed at GG/IVL, using algorithms that are designed for automatic malaria diagnosis, without user input. Versions of a prototype of the device were first tested in field settings in Thailand in 2014-2015 at clinics operated by the Shoklo Malaria Research Unit (SMRU) and then again in 2016-2017. When compared to expert microscopy at SMRU, the performance of the device with respect to diagnostic sensitivity (87.8%), species identification (85.6% species correctly identified) and parasite density estimation (44% of estimates within +/-25% of reference microscopy result) corresponded to WHO Competence Level 2. The device and the accompanying image analysis algorithms have since been further developed and a new, third version of the prototype is now available for testing in diverse settings with varying malaria prevalence and user expertise.

DETAILED DESCRIPTION:
The primary purpose of this evaluation is to quantify the diagnostic performance of the EasyScan Go prototype in various field settings. The performance of the EasyScan Go prototype will be assessed by scanning of negative and positive slides with the EasyScan Go and comparing the results with expert microscopy. Plasmodium genus- and species-specific PCR will also be performed on samples collected at some sites as an additional confirmatory test for the detection of malaria parasites and their species if present. Testing by microscopy and EasyScan Go will be performed in field clinic settings on Giemsa-stained slides prepared from febrile patient blood collected from a finger-prick. Further work will be undertaken at the WWARN laboratory in Bangkok for data analyses and for quality assurance.

Funder: Intellectual Ventures Lab/Global Good (2018) Sponser: University of Oxford Grant refernce number:The Global Good Fund I, LLC PA No.5

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age ≥ 6 months to 75 years
* Febrile at presentation or history of fever in the past 48 hours (≥ 37.5 ºC) and no other obvious diagnosis or cause for fever, warranting malaria investigation under routine clinical practice.
* Individual informed assent/consent obtained

Exclusion Criteria:

- Signs of severe malaria as defined by WHO

Ages: 6 Months to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The multi-centric evaluation is currently planned for implementation at relatively few sites/countries and the primary criteria for the selection of sites will be based on operational feasibility of the project, i.e., availability of resources to perform the study procedures, adequate expected numbers of malaria positive cases, etc.
  Potential sites in Senegal, Kenya, Tanzania, Uganda, Congo, South Africa, Burkina Faso, Brazil, Thailand, Indonesia, Bangladesh, Myanmar and Cambodia are being considered for the study.
  A minimum of 80 malaria cases confirmed by expert microscopy and a minimum of 80 malaria-negative cases per study site.
Sampling Method: Probability Sample
Enrollment: 2250 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity for malaria parasite detection | 6 months
Diagnostic specificity for malaria parasite detection | 6 months
Kappa statistic for parasite species identification | 6 months
Bland-Altman plots for parasite density estimation | 6 months

SECONDARY OUTCOMES:
Reliability (comparison between 2 devices and repeat reads) | 6 months
Cost-effectiveness as compared with routine methods | 6 months
Prevalence of parasite genetic markers of resistance to antimalarials by location and time period | 6 months
Prevalence of parasites carrying deletions of pfhrp2/3 genes by location and time period | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Das D, Vongpromek R, Assawariyathipat T, Srinamon K, Kennon K, Stepniewska K, Ghose A, Sayeed AA, Faiz MA, Netto RLA, Siqueira A, Yerbanga SR, Ouedraogo JB, Callery JJ, Peto TJ, Tripura R, Koukouikila-Koussounda F, Ntoumi F, Ong'echa JM, Ogutu B, Ghimire P, Marfurt J, Ley B, Seck A, Ndiaye M, Moodley B, Sun LM, Archasuksan L, Proux S, Nsobya SL, Rosenthal PJ, Horning MP, McGuire SK, Mehanian C, Burkot S, Delahunt CB, Bachman C, Price RN, Dondorp AM, Chappuis F, Guerin PJ, Dhorda M. Field evaluation of the diagnostic performance of EasyScan GO: a digital malaria microscopy device based on machine-learning. Malar J. 2022 Apr 12;21(1):122. doi: 10.1186/s12936-022-04146-1. PMID 35413904